CLINICAL TRIAL: NCT03020056
Title: Impact of Cataract Surgery to Socioeconomic Status in Rural Area of Southern China: A Randomised Controlled Trial
Brief Title: Impact of Cataract Surgery to Socioeconomic Status in Rural Area
Acronym: ICSSES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhi Liu, Clinical Professor,director of Zhongshan Ophthalmic Center, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016KYYJ007
Record Dates: First submitted 2016-11-26; First posted 2017-01-13 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Cataract Surgery
Keywords: cataract surgery; socioeconomic status; quality of life; rural area; China; randomized controlled trial
MeSH Terms: interventions — Cataract Extraction; Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- waiting surgery (Placebo Comparator): Cataract surgery will be performed at 1 year after enrollment.These participants will be provided with Phacolin eye drops(Zhongshan ophthalmic center, China).
  Interventions: Drug: Phacolin eye drops
- expedited surgery (Experimental): Cataract surgery will be performed within 4 weeks.
  Interventions: Procedure: cataract surgery

INTERVENTIONS:
Drug: Phacolin eye drops — After enrollment, the participants will be provided antioxidant eye drops, Phacolin (Zhongshan ophthalmic center, China) for free.The eye drops will be administered 4 times per day for 1 year.Then either phacoemulsification or manual small incision cataract surgery will be performed.
  Other Names: antioxidant eye drops
  Arms: waiting surgery
Procedure: cataract surgery — After enrollment,either phacoemulsification or manual small incision cataract surgery will be performed within 4 weeks.
  Other Names: phacoemulsification or MSICS
  Arms: expedited surgery

SUMMARY:
This is a randomized controlled trial to investigate the effect of cataract surgery on the socioeconomic status of cataract patients in rural area of Southern China.

DETAILED DESCRIPTION:
Cataract is the leading cause of visual impairment worldwide and surgery is the only effective treatment. Previous studies show that visual impairment impacts the patient's socioeconomic status(SES). However, how cataract surgery affects the SES of cataract patients in rural area of China has not been determined before.

In the investigators study, cataract patients in rural area of Southern China will be enrolled and randomly divided into two groups. Cataract surgery will be performed in 4 weeks in intervention group, while performed at 1 year later in control group. The annual personal income by work, annual household income, hours in paid and unpaid work in the previous month, real estate ownership, household expenditures and quality of life will be investigated before and 1 year after surgery. Then, the difference in SES and quality of life change between two groups at 1 year later will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract patients aged over 50 with best corrected visual acuity (BCVA) less than 0.3 in the better eye.

Exclusion Criteria:

* History of other eye disease that contributes to visual impairment, including keratopathy, uveitis, glaucoma, retinopathy, ocular trauma, or intraocular surgery.
* Cases in need of expedited surgery, including shallow anterior chamber (central anterior chamber depth less than 2 mm and/or peripheral anterior chamber depth less than 1/4 corneal thickness), blindness of grade IV and V (BCVA less than 0.02 in the better eye), and intumescent or hypermature stage of cortical cataract.
* Systemic disease dampening activity, including cardiovascular and cerebrovascular diseases, hemiplegia, neurodegenerative diseases such as Alzheimer's disease and Parkinson's disease.
* Patients not willing to participate in the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
annual personal income by work in Chinese Yuan | 1 year
  The annual personal income comprises of the direct and the indirect income by work. The indirect income is derived from unpaid work and calculated as follows: unpaid work time × local income per hour.

SECONDARY OUTCOMES:
Health-related quality of life score | 1 year
  Health-related QoL score will be measured by EuroQol 5 dimensions with 5 levels (EQ-5D-5L) and self-rated health (SRH). For each dimension, participants are asked to mark between 1: "no problems" to 5: "unable to/extreme problems". Self-rated health using a vertical Visual Analogue Scale (VAS), with scores ranging from 0 (representing worst imaginable health state) to 100 (best imaginable health state).
  1. mobility
  2. self-care
  3. usual activities
  4. pain/discomfort
  5. anxiety/depression f: self-rated health
Vision related quality of life score | 1 year
  Vision related QoL score will be measured by Catquest-9S, which is a short form of Catquest questionnaire. The Catquest-9SF questionnaire comprises 7 questions for performing daily-life activities and 2 global questions about difficulties in general and satisfaction with vision (1= very great difficulty; 2= great difficulty; 3= some difficulty; 4= no difficulty).
  1. reading text in the newspaper
  2. recognizing faces of people you meet
  3. seeing prices of goods when shopping
  4. seeing to walk on uneven ground
  5. seeing to do needlework and handicraft
  6. reading text on television
  7. seeing to carry out a preferred hobby
  8. difficulty in daily life
  9. satisfaction on present vision

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, Doctor, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Yingfeng Zheng, Doctor, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Huidong people's hospital, Huidong, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tan X, Han X, Zheng Y, Jin L, Qiu X, Zhu Y, Chen C, Zhang J, Dickey H, Wang D, Huang S, Liu B, Liang X, Zeng Y, Lin H, He M, Luo L, Huang W, Congdon N, Liu Y. Impact of Cataract Surgery on Income in Rural Southern China: The SUCCESS Randomized Controlled Trial. Asia Pac J Ophthalmol (Phila). 2023 Jul-Aug 01;12(4):355-363. doi: 10.1097/APO.0000000000000624. Epub 2023 Jul 21. PMID 37523426